CLINICAL TRIAL: NCT05603962
Title: The Effectiveness of Visual Training Using Prisms on Visual Symptoms and Binocular Vision in Convergence Insufficiency Patients
Brief Title: The Effectiveness of Visual Training in Convergence Insufficiency Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202207058RINB
Record Dates: First submitted 2022-10-25; First posted 2022-11-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-03

CONDITIONS: Convergence Insufficiency
Keywords: Visual training; Prism; Binocular vision
MeSH Terms: conditions — Ocular Motility Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop training group (Active Comparator): Home-base prism training during week 1-6 --> then stop training during week 7-12 --> endpoint data collected at week 12
  Interventions: Behavioral: Visual training
- Continune training group (Experimental): Home-base prism training during week 1-12 --> endpoint data collected at week 12
  Interventions: Behavioral: Visual training

INTERVENTIONS:
Behavioral: Visual training — Visual training is the main type of management for CI patients clinically; however, the existing training protocol required patients to make several visits to the clinic for visual training, which might increase the burden for patients and result in higher failures in training. Therefore, this study will use a simple training method by utilizing prisms for CI patients to train at home, then compare visual symptoms and binocular vision after the training.

SUMMARY:
Convergence insufficiency (CI) is one of the most common binocular vision disorders. The prevalence of CI ranges from 3% to 6% in school-aged children. CI symptoms include visual fatigue, headache, blurred vision, and diplopia and could be caused while using near-distance viewing. These symptoms might become more severe with increasing need to perform near-distance tasks. Long-term visual symptoms could result in a negative impact on learning behaviors and work performance in patients. Nowadays, visual training is the main type of management for CI patients clinically; however, the existing training protocol required patients to make several visits to the clinic for visual training, which might increase the burden for patients and result in higher failures in training. Therefore, this study will use a simple training method by utilizing prisms for CI patients to train at home, then compare visual symptoms and binocular vision after the training. In stage I of this study, investigators will recruit 60 symptomatic CI participants aged 9 to 30 years old to do a 6-week visual training with the prisms (15 min/time, 3 times/week). The post-training outcomes will be collected at week 4 and week 6. In stage II, all of the participants will be randomly divided into the "stop training group" and the "continue training group." The participants in the "continue training group" will have the same 6-week prism training and in the "stop training group" will stop all the prism training during this period. The final post-training outcomes of all the participants will be collected again at week 12. In this study, investigators will investigate the effectiveness of the prisms training for 6 weeks and for 12 weeks on visual symptoms and binocular vision in CI patients, and evaluate whether the training effect will be affected by stopping training after 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The overall score of CI symptom survey ≥ 16 (9-18 years old) or ≥ 21 (19-30 years old)
2. The break point of near point of convergence (NPC) ≥ 6 cm
3. Exophoria at near distances be at least 4∆ higher than at far distances
4. Near positive fusional vergence (PFV) ≤ 15∆ or failing Sheard's criterion at near.

Exclusion Criteria:

1. The best corrected visual acuity (BCVA) of < 20/25 in each eye at far and near distances
2. Amblyopia patients or the difference of BCVA between the two eyes ≥ 2 lines
3. Constant strabismus patients
4. History of strabismus surgery or refractive surgery
5. Systemic diseases that would affect binocular vision
6. Acquired brain injury or neurological disorder.

Ages: 9 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Binocular vision and visual function evaluation | 12 weeks for each participant
  Change from baseline best corrected visual acuity: distance visual acuity measured for each eye at a distance of 6 m and at near 40 cm for each eye will be measured using Snellen charts. NPC and the amplitude of accommodation will be measured using Royal Air Force (RAF) rule. Stereoacuity will be measured by the Random dot stereotest.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Hsun Tsai, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei County, Taiwan